CLINICAL TRIAL: NCT01096186
Title: An Open Label Extension Study of the Safety and Clinical Utility of IPX066 in Subjects With Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPX066-B09-03
Record Dates: First submitted 2010-03-25; First posted 2010-03-31 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2017-01

CONDITIONS: Parkinson's Disease
Keywords: motor Symptoms; efficacy; IPX066; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label IPX066 (Other): Subjects received IPX066 95 mg, IPX066 145 mg, IPX066 195 mg, or IPX066 245 mg for approximately 9 months. The dose and dosing frequency was determined by the investigator.
  Interventions: Drug: IPX066 95 mg; Drug: IPX066 145 mg; Drug: IPX066 195 mg; Drug: IPX066 245 mg

INTERVENTIONS:
Drug: IPX066 95 mg — 23.75 - 95 mg CD-LD capsules
  Other Names: CD-LD ER 95 mg
Drug: IPX066 145 mg — 36.25 - 145 mg CD-LD capsules
  Other Names: CD-LD ER 145 mg
Drug: IPX066 195 mg — 48.75 - 195 mg CD-LD capsules
  Other Names: CD-LD ER195 mg
Drug: IPX066 245 mg — 61.25 - 245 mg CD-LD capsules
  Other Names: CD-LD ER 245 mg

SUMMARY:
The purpose of this study is to determine the long term safety and clinical utility of IPX066 in subjects with Parkinson's Disease.

DETAILED DESCRIPTION:
IPX066 is intended for chronic treatment of motor symptoms for all stages of PD. This study is designed to enroll subjects who have successfully completed one of the following studies of IPX066:

* IPX066-B08-05 (A Placebo-Controlled Study to Evaluate the Safety and Efficacy of IPX066 in Subjects with Parkinson's Disease)
* IPX066-B08-11 (A Study to Compare Pharmacokinetics and Pharmacodynamics of IPX066 to Standard Carbidopa - Levodopa)
* IPX066-B09-02 (A Study to Evaluate the Safety and Efficacy of IPX066 in Advanced Parkinson's Disease)

All participants will be given IPX066 for 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must meet the following inclusion criteria in order to be enrolled in the study:

  1. Successful completion of studies IPX066-B08-05, IPX066-B08-11, or IPX066-B09-02.
  2. In the opinion of the Investigator, the Parkinson's disease diagnosis is still valid and the subject remains eligible for LD therapy.

Exclusion Criteria:

* Each subject must be free of the following exclusion criteria in order to be enrolled in the study:

  1. Received an investigational medication other than those from an IPX066 trial within 4 weeks prior to the planned start of treatment.
  2. Anticipates functional neurosurgical treatment for PD (e.g., ablation or deep brain stimulation) during study participation.
  3. Received within 4 weeks prior to Baseline Visit or planning to take during study participation: nonselective monoamine oxidase (MAO) inhibitors (with the exception of rasagiline).
  4. In the opinion of the Investigator, should not participate in the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (81):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mohammed Ali Parkinson's Center, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Clinical Trials Inc., Little Rock, Arkansas
  - Coastal Neurological Medical Group, La Jolla, California
  - Coordinated Clinical Research, La Jolla, California
  - The Parkinson's Institute, Sunnyvale, California
  - Collaborative NeuroScience Network, Inc., Torrance, California
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Sunrise Clinical Research, Hollywood, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charlotte Neurological Services Parkinson's Disease Treatment Center of S.W. Florida, Port Charlotte, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - University of South Florida, Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Medical College of Georgia, Movements Disorders Clinic, Augusta, Georgia
  - Movement Disorder Center at Idaho Elks Rehabilitation Hospital, Boise, Idaho
  - Northwestern University, Feinberg School of Medicine, Dept. of Neurology, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Quest Research Institute, Bingham Farms, Michigan
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - UMDNJ Robert Wood Johnson Medical Center, Department of Neurology, New Brunswick, New Jersey
  - Albany Medical College, Parkinson's Disease and Movement Disorders Center, Albany, New York
  - David L. Kreitzman, MD, P.C., Commack, New York
  - Columbia University Neurological Institute, New York, New York
  - Institute for Human Performance, Syracuse, New York
  - Duke University Medical Center Movement Disorders Center, Durham, North Carolina
  - University Neurology, Inc., Cincinnati, Ohio
  - University of Toledo, Toledo, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - South Puget Sound Neurology, Tacoma, Washington
  - Wisconsin Institute for Neurologic and Sleep Disorders, Milwaukee, Wisconsin
- Canada (4):
  - London Health Sciences Centre, University Hospital, London, Ontario
  - Parkinson's & Neurodegenerative Disorder Clinic, Ottawa, Ontario
  - Ottawa Hospital Civic Site, Ottawa, Ontario
  - Quebec Memory & Motor Skills Disorders Clinic, Québec, Quebec
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - West Tallinn Central Hospital,, Tallinn
- Germany (3):
  - Praxis für Neurologie und Psychiatrie, Westerstede, Lower Saxony
  - Neurozentrm - Praxis fur Neurologie und Psychiatrie, Berlin
  - Neurologiepraxis, Berlin
- Latvia (2):
  - P.Stradina university hospital, Riga
  - Gailezers hospital, Riga
- Lithuania (5):
  - Kaunas Medical University Hospital, Kaunas
  - Siauliai Regional Hospital, Šiauliai
  - National Centre of Osteoporosis, Vilnius
  - Vilnius University Emergency Hospital, Vilnius
  - Vilnius University Hospital Santariskiu klinikos, Vilnius
- Poland (7):
  - PALLMED Sp. z o.o., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Krakowska Akademia Neurologii Sp. z o. o., Krakow, Lesser Poland Voivodeship
  - Wojewódzki Szpital Specjalistyczny im. Stefana Kardynala Wyszynskiego, SPZOZ w Lublinie, Lublin, Lublin Voivodeship
  - Centrum Leczenia Chorób Cywilizacyjnych Sp. z o. o. S. K. A., Warsaw, Masovian Voivodeship
  - Euromedis Sp. z o.o., Szczecin, West Pomeranian Voivodeship
  - Gabinet Neurologiczny, Indywidualna Specjalistyczna Praktyka Lekarska, Mosina, Wielkopoloskie
  - Neuro-Care NZOZ, Katowice
- Romania (8):
  - Clinical Rehabilitation Hospital Iasi, Neurology Department, Lasi, Romania
  - Psychiatry and Neurology Hospital Brasov, Neurology Department, Brasov
  - Neomed Research, Brasov
  - Colentina Clinical Hospital Bucharest, II Neurology Department, Bucharest
  - CFR Clinical Hospital Constanta, Neurology Department, Constanța
  - County Clinical Emergency Hospital Targu Mures, I Neurology Department, Târgu Mureş
  - County Clinical Emergency Hospital Targu Mures, II Neurology Department, Târgu Mureş
  - County Clinical Emergency Hospital Timisoara, Neurology Department, Timișoara
- Spain (2):
  - Hospital General de Cataluña, Sant Cugat del Vallès, Barcelona
  - Clinica Ruber SA, Madrid
- Ukraine (12):
  - Department of neurology and neurosurgery of Dnipropetrovsk State Medical Academy based on Dnipropetrovsk regional hospital named after Mechnikov, Dnipropetrovsk
  - Department of Psychiatry and Medical Psychology of Donetsk National Medical University, Donetsk
  - Department of Neurological Diseases and Medical Genetic of Donetsk National Medical University, Donetsk
  - 1st neurology department of Central Clinical Hospital of Ukrzaliznytsya, Kharkiv
  - Department of Vascular Pathology of brain of Institute of neurology, psychiatry and narcology of AMS of Ukraine, Kharkiv
  - Institute of Neurology, Psychiatry and Narcology of the AMS of Ukraine, Kharkiv
  - Neurology department of Lviv regional clinical hospital, Lviv
  - Odessa Regional Clinical Hospital, Dept. of Neurosurgery, Odesa
  - Neurology department of Medical Dental Academy based on Poltava regional hospital, Poltava
  - Vinnytsia Regional Psycho-Neurological Hospital, Vinnytsia
  - Zaporizhzhya State Medical University based at Zaporizhzhya State Clinical Hospital #6, Zaporizhzhya
  - Zaporozhye Regional Clinical Hospital, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study dates March 25, 2010 through October 19, 2011 Completion of previous trial a requirement
Groups:
- IPX066: Open-label IPX066 Dose was individualized for each subject in the study. IPX066 doses could be adjusted throughout the study.
Period: Overall Study
Arm/Group | IPX066
Started | 617
Completed | 567
Not Completed | 50
Not completed — Adverse Event | 16
Not completed — Death | 4
Not completed — Lack of Efficacy | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 22
Not completed — Physician Decision | 1
Not completed — Noncompliance with study drug | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Arm/Group | IPX066
Number analyzed (Participants) | 617
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234
  Male | 383
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 582
  Unknown or Not Reported | 15
Race/Ethnicity, Customized [Number; unit: participants]
  White | 608
  Black or African American | 3
  Asian | 3
  Other | 3
Region of Enrollment [Number; unit: participants]
  Canada | 48
  Latvia | 2
  Romania | 43
  United States | 260
  Ukraine | 165
  Poland | 50
  Lithuania | 18
  Germany | 19
  Estonia | 3
  Spain | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Sum of UPDRS Part II + UPDRS Part III
Description: Analysis of the Change from Baseline in the sum of the Unified Parkinson's Disease Rating Scale (UPDRS) Part II (Activities of Daily Living) + UPDRS Part III (Motor Examination) at End of Study.
  Unified Parkinson's Disease Rating Scale (UPDRS) - Four Parts Higher score values represent a worse outcome.
  Subscales II and III were summed:
  Part I: Mentation, Behavior and Mood - 4 questions 1-4 Score range: 1-16 Part II: Activities of Daily Living - 13 questions 5-17 Score range: 0-52 Part III: Motor Examination - 19 questions 18-31 and 25 total assessments Score range: 0-100 Part IV: Complications of Therapy (In the past week) - 11 questions Score range: 0-25
Time Frame: 9 months
Population: All enrolled subjects with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IPX066
Number analyzed (Participants) | 567
units on a scale | 26.4 (13.3)

2. Secondary Outcome: Total UPDRS Parts I-IV
Description: Analysis of the Change from Baseline in the sum of the Unified Parkinson's Disease Rating Scale (UPDRS) Part I (Mentation, Behavior and Mood), Part II (Activities of Daily Living), UPDRS Part III (Motor Examination), and Part IV (Complications of Therapy [In the past week]) at End of Study. Includes both scoring by a clinician and a historical report of mental functioning, activities of daily living and complications of therapy in the past week obtained by questioning the patient.
  Unified Parkinson's Disease Rating Scale (UPDRS) - Four Parts Higher score values represent a worse outcome.
  Subscales II and III were summed:
  Part I: Mentation, Behavior and Mood - 4 questions 1-4 Score range: 1-16 Part II: Activities of Daily Living - 13 questions 5-17 Score range: 0-52 Part III: Motor Examination - 19 questions 18-31 and 25 total assessments Score range: 0-100 Part IV: Complications of Therapy (In the past week) - 11 questions Score range: 0-25
Time Frame: 9 months
Population: All enrolled subjects with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IPX066
Number analyzed (Participants) | 567
units on a scale | 30.5 (14.67)

3. Secondary Outcome: Patient Global Impression (PGI)
Description: Satisfaction of IPX066 using Patient Global Impression (PGI) 7-point scale.
  Patient Global Impression 0-7 - higher value indicates increased improvement from study start
Time Frame: 9 months
Population: All enrolled subjects with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IPX066
Number analyzed (Participants) | 567
units on a scale | 5.4 (1.16)

ADVERSE EVENTS:
Time Frame: Screening through 9 months
Arm/Group | IPX066
Serious Adverse Events (participants affected / at risk) | 43/617
Other Adverse Events (participants affected / at risk) | 122/617
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IPX066 (N=617)
Atrial fibrillation (Cardiac disorders) | 2
Atrioventricular block complete (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 3
Femur facture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Scalpula fracture (Injury, poisoning and procedural complications) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Freezing phenomenon (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
IIIrd nerve paralysis (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Paranoia (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pelvic prolapse (Reproductive system and breast disorders) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Toe operation (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IPX066 (N=617)
Insomnia (Psychiatric disorders) | 36
Fall (Injury, poisoning and procedural complications) | 33
Dyskinesia (Nervous system disorders) | 34
Nausea (Gastrointestinal disorders) | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results of the Study conducted at the Site shall not be made before the first multi-site publication by Sponsor.